CLINICAL TRIAL: NCT00586586
Title: Assessment and Treatment - Anxiety in Children and Adults (Child Part)
Brief Title: Effectiveness Study of CBT for Anxiety in Children
Acronym: ATACA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17563
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Separation Anxiety Disorder; Social Anxiety Disorder; Generalized Anxiety Disorder
MeSH Terms: conditions — Anxiety, Separation; Phobia, Social; Generalized Anxiety Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group CBT (Experimental): The behavioral intervention FRIENDS (cognitive behavior therapy program developed by P. Barratt) delivered in groups of 4 to 8. 10 weekly sessions plus 2 booster sessions.
  Interventions: Behavioral: Cognitive behavioural therapy
- Individual CBT (Experimental): The behavioral intervention FRIENDS (cognitive behavior therapy program developed by P. Barratt) delivered individually.
  10 weekly sessions plus 2 booster sessions.
  Interventions: Behavioral: Cognitive behavioural therapy
- Wait-list control (No Intervention): Wait-list control condition for 5 weeks after last child has been included.

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy — The FRIENDS program developed by Paula Barrett, 10 weekly sessions of 60-90 minutes, with two additional parent meetings, and booster sessions 4 and 12 weeks after treatment.
  Other Names: FRIENDS
  Arms: Group CBT; Individual CBT

SUMMARY:
The study aims to evaluate the effectiveness of a cognitive behaviour therapy program (FRIENDS) for anxiety disorders in children aged 8-15 years who have been referred to child and adolescent mental health clinics in Western Norway.

DETAILED DESCRIPTION:
Cognitive behaviour therapy (CBT) has been shown to be an efficacious treatment for anxiety disorders in youths when delivered in university settings. However, there is a lack of studies evaluating the effectiveness of CBT in regular clinical settings.

The current study will compare a CBT program developed for anxiety in youths (the FRIENDS program by Paula Barrett, Australia), with a wait-list control condition. Group and individual treatment will also be compared in the study. Groups will be divided by age, with younger including 8-12-year-olds, and older 12-15-year-olds. Parents are also involved at the end of all therapy sessions, as well as in separate parent sessions. Assessment and treatment is delivered by clinicians working in seven outpatient clinics in Western Norway.

There will be 10 therapy sessions, with booster sessions 4 and 12 weeks later. Effectiveness will be evaluated post-treatment, and at 1 and 5 years follow-up. The study will have a randomized design. Children randomized to the wait-list condition will be offered treatment if they still meet inclusion criteria after the waiting period.

ELIGIBILITY:
Inclusion Criteria:

* Meeting DSM-IV criteria for separation anxiety, social anxiety or generalized anxiety disorder based on the ADIS interview schedule

Exclusion Criteria:

* Pervasive developmental disorders, Selective mutism, Mental retardation
* Having severe obsessional/compulsive, conduct or language problems.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2008-01-02; Primary Completion 2012-06-01 (Actual); Study Completion 2014-03-21 (Actual)

PRIMARY OUTCOMES:
Anxiety disorders according to the ADIS-IV C/P interview | Post-treatment and 1 and 5 year follow-up
  Diagnostic recovery from inclusion diagnoses and reduction on the clinical severity scale.

SECONDARY OUTCOMES:
Anxiety symptom score according to the Spence Children Anxiety Scale | Post-treatment, 1 and 5 year follow-up
Depressive symptoms according to the Mood and Feelings Questionnaire | Post-treatment, 1 and 5 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Einar Heiervang, MD, Principal Investigator — Haukeland University Hospital; Gro Janne H Wergeland, MD PhD, Study Chair — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Result] Wergeland GJ, Fjermestad KW, Marin CE, Haugland BS, Bjaastad JF, Oeding K, Bjelland I, Silverman WK, Ost LG, Havik OE, Heiervang ER. An effectiveness study of individual vs. group cognitive behavioral therapy for anxiety disorders in youth. Behav Res Ther. 2014 Jun;57:1-12. doi: 10.1016/j.brat.2014.03.007. Epub 2014 Mar 31. PMID 24727078
- [Result] Wergeland GJ, Fjermestad KW, Marin CE, Haugland BS, Silverman WK, Ost LG, Havik OE, Heiervang ER. Predictors of dropout from community clinic child CBT for anxiety disorders. J Anxiety Disord. 2015 Apr;31:1-10. doi: 10.1016/j.janxdis.2015.01.004. Epub 2015 Jan 22. PMID 25637909
- [Result] Wergeland GJ, Fjermestad KW, Marin CE, Bjelland I, Haugland BS, Silverman WK, Ost LG, Bjaastad JF, Oeding K, Havik OE, Heiervang ER. Predictors of treatment outcome in an effectiveness trial of cognitive behavioral therapy for children with anxiety disorders. Behav Res Ther. 2016 Jan;76:1-12. doi: 10.1016/j.brat.2015.11.001. Epub 2015 Nov 5. PMID 26583954
- [Derived] Kodal A, Fjermestad K, Bjelland I, Gjestad R, Ost LG, Bjaastad JF, Haugland BSM, Havik OE, Heiervang E, Wergeland GJ. Long-term effectiveness of cognitive behavioral therapy for youth with anxiety disorders. J Anxiety Disord. 2018 Jan;53:58-67. doi: 10.1016/j.janxdis.2017.11.003. Epub 2017 Nov 26. PMID 29195188
- [Derived] Fjermestad KW, Lerner MD, McLeod BD, Wergeland GJ, Heiervang ER, Silverman WK, Ost LG, De Los Reyes A, Havik OE, Haugland BS. Therapist-youth agreement on alliance change predicts long-term outcome in CBT for anxiety disorders. J Child Psychol Psychiatry. 2016 May;57(5):625-32. doi: 10.1111/jcpp.12485. Epub 2015 Dec 9. PMID 26647901